CLINICAL TRIAL: NCT02835599
Title: Registry for the EVolution Of LUng Cancer Therapy Implementation and Outcomes Now
Acronym: REVOLUTION
Status: Terminated | Type: Observational
Why Stopped: The study sponsor requested the study be terminated as the existing study design did not meet their needs.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00110
Record Dates: First submitted 2016-07-08; First posted 2016-07-18 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Archived residual specimens will be requested from appropriate institution for each patient at consent. One block or 20 slides (if block is not available) will be requested for each patient for molecular testing and sent as directed by the Lab Manual. Specimens will be banked at the Carolinas HealthCare Biospecimen Repository (CHS BSR) specifically for this protocol in their Clinical Trials Management System Biospecimen Module (CTMS BSM).
Oversight: Data Monitoring Committee: No

SUMMARY:
REVOLUTION will be a US multicenter observational registry in scope and governed by a steering committee of approximately 8 experts in NSCLC and outcomes research. The primary goal of the registry is characterizing patterns of use for NSCLC therapy. REVOLUTION will be a multicenter registry enrolling approximately 2,500 patients. Additional patients limited to those with EGFR mutations may be enrolled following the initial study period as needed to ensure adequate sample sizes needed to examine primary questions of interest in the EGFR mutant population. Patients will be enrolled over a three year period across approximately 25 geographically diverse academic as well as community based sites within the US. The five year follow-up period will ensure robust survival data for correlations with clinical, tumor, and treatment variables.

The target of 2,500 patients is meant to ensure adequate numbers of NSCLC patients with particular characteristics of interest including patients with adenocarcinoma, and EGFR mutations and effectively evaluate these patients with respect to key outcomes of interest including overall survival, time to progression, stage at progression, secondary metastases including brain metastases (at diagnosis and progression), comorbidity burden, and performance status at index date.

The study design allows a cross-sectional perspective with collection of detailed patient and clinical characteristics at enrollment followed by longitudinal assessment of clinician and patient-reported endpoints every three months. Centralized follow-up will be conducted by having sites upload patient data following each visit via the web-based data system, with patients who do not show up for site visits being contacted via telephone by the Duke Clinical Research Institute (DCRI) call center. Site recruitment and patient enrollment will be weighted based upon provider specialty and ability to enroll patients with NSCLC with the specified inclusion criteria.

DETAILED DESCRIPTION:
REVOLUTION will be a US multicenter observational registry in scope and governed by a steering committee of approximately 8 experts in NSCLC and outcomes research. The primary goal of the registry is characterizing patterns of use for NSCLC therapy. REVOLUTION will be a multicenter registry enrolling approximately 2,500 patients. Additional patients limited to those with EGFR mutations may be enrolled following the initial study period as needed to ensure adequate sample sizes needed to examine primary questions of interest in the EGFR mutant population. Patients will be enrolled over a three year period across approximately 25 geographically diverse academic as well as community based sites within the US. The five year follow-up period will ensure robust survival data for correlations with clinical, tumor, and treatment variables.

The target of 2,500 patients is meant to ensure adequate numbers of NSCLC patients with particular characteristics of interest including patients with adenocarcinoma, and EGFR mutations and effectively evaluate these patients with respect to key outcomes of interest including overall survival, time to progression, stage at progression, secondary metastases including brain metastases (at diagnosis and progression), comorbidity burden, and performance status at index date.

The study design allows a cross-sectional perspective with collection of detailed patient and clinical characteristics at enrollment followed by longitudinal assessment of clinician and patient-reported endpoints every three months. Centralized follow-up will be conducted by having sites upload patient data following each visit via the web-based data system, with patients who do not show up for site visits being contacted via telephone by the Duke Clinical Research Institute (DCRI) call center. Site recruitment and patient enrollment will be weighted based upon provider specialty and ability to enroll patients with NSCLC with the specified inclusion criteria.

Study Patient Selection Criteria

Patients are eligible to be included in the study if they meet all of the following criteria:

1. ≥19 years of age
2. Patients with a primary diagnosis of NSCLC within the past 5 years who are eligible for their first systemic therapy based on disease characteristics. Systemic therapy may include any cytotoxic, targeted, immune-based, or otherwise non-local treatment modality. Specific allowed settings include the following:

   * Incident metastatic disease (stage IV) undergoing palliative therapy
   * Non-metastatic disease undergoing adjuvant, neoadjuvant, or concurrent chemoradiation with either curative or palliative intent
   * Recurrent or subsequently metastatic disease (any stage)
3. Pathologic confirmation of malignancy prior to initiation of first systemic therapy
4. Patient agrees to the submission of archival biospecimen sample(s) (collected up to two years prior) for analysis
5. Availability of key variables at the time of screening (e.g. stage, demographics)
6. Have been fully informed and are able to provide written consent for longitudinal follow-up and agree to be accessible by phone
7. Patients may be concurrently enrolled in unblinded clinical trials, but not blinded clinical trials in which the treatment being administered is unknown

Patients are excluded if they meet any of the following criteria:

1. Pre-specified enrollment caps have been met (Figure 1)
2. Suspected recurrent or subsequently metastatic disease that is not biopsy confirmed prior to receipt of initial systemic therapy

ELIGIBILITY:
Inclusion Criteria:

1. ≥19 years of age
2. Patients with a primary diagnosis of NSCLC within the past 5 years who are eligible for their first systemic therapy based on disease characteristics. Systemic therapy may include any cytotoxic, targeted, immune-based, or otherwise non-local treatment modality. Specific allowed settings include the following:

   1. Incident metastatic disease (stage IV) undergoing palliative therapy
   2. Non-metastatic disease undergoing adjuvant, neoadjuvant, or concurrent chemoradiation with either curative or palliative intent
   3. Recurrent or subsequently metastatic disease (any stage)
3. Pathologic confirmation of malignancy prior to initiation of first systemic therapy
4. Submission of archival biospecimen sample(s) (collected up to two years prior) for analysis
5. Availability of key variables at the time of screening (e.g. stage, demographics)
6. Have been fully informed and are able to provide written consent for longitudinal follow-up and agree to be accessible by phone
7. Patients may be concurrently enrolled in unblinded clinical trials, but not blinded clinical trials in which the treatment being administered is unknown

Exclusion Criteria:

1. Pre-specified enrollment caps have been met (Figure 1)
2. Suspected recurrent or subsequently metastatic disease that is not biopsy confirmed prior to receipt of initial systemic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be enrolled over a three year period across approximately 25 geographically diverse academic as well as community based sites within the US. The five year follow-up period will ensure robust survival data for correlations with clinical, tumor, and treatment variables.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment decisions using molecular testing and results, provider decisions and patient preferences. | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Characterize current practice patterns for the care of patients with NSCLC, with a special emphasis on pharmacotherapy (i.e. chemotherapy, targeted agents, and immunotherapy) and patients with EGFR mutated disease. These data will include treatment, molecular test administration and results, provider decisions and patient preferences, and explore the determinants of each.
Assessment of progression-free survival | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Compare progression-free survival, overall survival, and duration of response associated with targeted therapies, immune checkpoint inhibitors, and cytotoxic chemotherapy in NSCLC and EGFR mutated disease.
Assessment of overall survival | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Compare progression-free survival, overall survival, and duration of response associated with targeted therapies, immune checkpoint inhibitors, and cytotoxic chemotherapy in NSCLC and EGFR mutated disease.
Assessment of treatments. | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Compare of progression-free survival, overall survival, and duration of response associated with targeted therapies, immune checkpoint inhibitors, and cytotoxic chemotherapy in NSCLC and EGFR mutated disease.

SECONDARY OUTCOMES:
Assessment of billing claims data. | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assessments will be aggregated to quantify total, treatment-related, and toxicity-related health care resource utilization and associated financial burden at the population level (not at the individual patient level) using a three-pronged approach including 1) costs extracted from site billing claims, 2) payments obtained from Medicare claims and 3) both objective and subjective measures of patient financial burden to be collected alongside PROs.
Assessment of patient demographics, smoking history and disease characteristics | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Characterize the current landscape of actionable mutations in the general clinical population and identify additional factors such as demographics, smoking history, and disease characteristics that predict the presence of actionable mutations as well as the development of T790M mutations in patients with EGFR mutated disease at initial presentation.
Assessment of patient hospitalizations. | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assess quality of life (QOL) associated with various treatment regimens and the association of severe complications (i.e. hospitalizations, emergency room visits) with treatment.
Assessment of targeted, immune, and cytotoxic therapies | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assess patient reported outcomes associated with commonly used targeted, immune, and cytotoxic therapies and additionally measures of patient reported objective and subjective financial burden as a result of their cancer treatment.
Assessment of financial burden related to treatment | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assess patient reported outcomes associated with commonly used targeted, immune, and cytotoxic therapies and additionally measures of patient reported objective and subjective financial burden as a result of their cancer treatment.
Assessment of EGFR mutation status. | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Characterize and describe the NSCLC patient population as a whole and by EGFR mutation status, with emphasis on demographics and comorbidities.
Assessment of molecular markers using tissue specimens. | Time from first patient enrolled up to study completion, approximately 3 years.
  Bank archived tissue specimens for future assessment of molecular markers identified in this or other relevant studies.
Assessment of molecular markers using blood specimens | Time from first patient enrolled up to study completion, approximately 3 years.
  Analyze other specimens (eg blood) for future assessment of molecular markers.
Assessment of costs extracted from site billing claims | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assessments will be aggregated to quantify total, treatment-related, and toxicity-related health care resource utilization and associated financial burden at the population level (not at the individual patient level) using a three-pronged approach including 1) costs extracted from site billing claims, 2) payments obtained from Medicare claims and 3) both objective and subjective measures of patient financial burden to be collected alongside PROs.
Assessment of patient financial burden using the Patient reported objective and subjective measures of financial toxicity patient questionnaire | Time from first patient enrolled to data cut of assessed approximately every 6 months up to 72 months.
  Assessments will be aggregated to quantify total, treatment-related, and toxicity-related health care resource utilization and associated financial burden at the population level (not at the individual patient level) using a three-pronged approach including 1) costs extracted from site billing claims, 2) payments obtained from Medicare claims and 3) both objective and subjective measures of patient financial burden to be collected alongside PROs.

OTHER OUTCOMES:
Assessment of patient treatments | Time from first patient enrolled up to 3 years.
  Generate empiric evidence to assess current NSCLC treatment paradigms with and without EGFR mutations, including combination therapy, and hypothesize rational alternative treatment sequences to optimize the care of patients treated in general clinical practice.
Evaluate multiple comorbidities and low socioeconomic status | Time from first patient enrolled up to 3 years
  Characterize patterns of care and outcomes in patients with aggressive disease and poor baseline health. Specifically, we will explore variation in the management and outcomes of patients with higher baseline health risk (i.e. multiple comorbidities, low socioeconomic status) as well as those who present with more advanced disease (e.g. multiple metastases, symptomatic disease, weight loss). Through completion of this objective we hope to help inform personalized risk-benefit assessment for patients whose management is challenging yet are not represented within most clinical trials.
Evaluate patients with advanced disease (e.g. multiple metastases, symptomatic disease, weight loss) | Time from first patient enrolled up to 3 years
  Characterize patterns of care and outcomes in patients with aggressive disease and poor baseline health. Specifically, we will explore variation in the management and outcomes of patients with higher baseline health risk (i.e. multiple comorbidities, low socioeconomic status) as well as those who present with more advanced disease (e.g. multiple metastases, symptomatic disease, weight loss). Through completion of this objective we hope to help inform personalized risk-benefit assessment for patients whose management is challenging yet are not represented within most clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Crawford, MD, Principal Investigator — Duke Clinical Research Institute; Edward Kim, MD, Study Chair — Atrium Health Levine Cancer Institute
Locations (15):
- United States (15):
  - Research Site, Monterey, California
  - Research Site, Santa Rosa, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Southfield, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Omaha, Nebraska
  - Research Site, Rock Hill, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Newport News, Virginia
  - Research Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Sponsor approval to share data is pending.

REFERENCES:
- See also: D133FR00110_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4095&filename=D133FR00110_FinalSummary_07.12.2017.pdf